CLINICAL TRIAL: NCT02439970
Title: SUSTAIN: A Randomized, Double-Blind, Multicenter, Phase 3 Study of the Efficacy, Safety, and Tolerability of Brincidofovir Versus Valganciclovir for the Prevention of Cytomegalovirus Disease in High-Risk Kidney Allograft Recipients
Brief Title: A Phase 3 Study of Brincidofovir Versus Valganciclovir for the Prevention of Cytomegalovirus Disease
Acronym: SUSTAIN
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated early due to results from another CMX001 study
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMX001-303
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Results first posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Cytomegalovirus Disease
Keywords: kidney transplant allograft; recipients
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — brincidofovir; Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment 1 (Active Comparator): 100 mg brincidofovir (BCV; 1 tablet) administered orally twice weekly, plus valganciclovir (vGCV) placebo (2 tablets) administered orally once daily.
  Interventions: Drug: Brincidofovir
- Treatment 2 (Active Comparator): 900 mg valganciclovir (vGCV; two 450 mg tablets) administered orally once daily, plus brincidofovir (BCV) placebo (1 tablet) administered orally twice weekly.
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Brincidofovir
  Other Names: CMX001; BCV
  Arms: Treatment 1
Drug: Valganciclovir
  Other Names: vGCV
  Arms: Treatment 2

SUMMARY:
To compare the efficacy of oral brincidofovir (BCV) to valganciclovir (vGCV) for the prevention of cytomegalovirus (CMV) disease in kidney transplant allograft recipients who are CMV seronegative pretransplant and received a kidney from a CMV seropositive donor

DETAILED DESCRIPTION:
This was a randomized, double-blind, double-dummy, parallel-group, multicenter study of the efficacy, safety, and tolerability of oral BCV versus vGCV for the prevention of CMV disease in high-risk kidney transplant allograft recipients, defined as CMV-seronegative recipients (R-) receiving a CMV-seropositive graft (D+). The study comprised a screening evaluation period (up to 14 days posttransplant), a treatment period (up to 28 weeks posttransplant), and a posttreatment follow-up period (24 weeks, through Week 52 posttransplant).

ELIGIBILITY:
Inclusion Criteria

Subjects must have met all of the following criteria, as applicable, to be eligible to participate in this study:

1. Were male or female kidney transplant recipients who were ≥18 years of age (subject to local law/practice for clinical trial participation) and ≤14 days following their first or second renal allograft.
2. Were at high risk of cytomegalovirus (CMV) infection defined as CMV-seronegative recipients who have received an allograft from a CMV-seropositive donor.
3. Had an estimated glomerular filtration rate of >10 mL/min (Cockcraft-Gault equation) at screening based on local laboratory results.
4. Were CMV viremia negative (i.e., "not detected") as measured by the desginated central virology laboratory using the Roche COBAS® AmpliPrep/COBAS® TaqMan® CMV Test no more than 5 days prior to subject randomization, and at all prior assessments performed since transplant under local standard of care.
5. Were able to ingest, absorb, and tolerate tablets.
6. If male, was willing to use an acceptable contraceptive method(s) throughout the duration of his participation in the study, i.e., through Week 52.
7. If female of childbearing potential, i.e., not post menopausal or surgically sterile, was willing to use 2 acceptable contraceptive methods, 1 of which must have been a barrier method, throughout the duration of her participation in the study, i.e., through Week 52.
8. Were willing and able to provide informed consent.
9. Were willing and able to participate in all required study activities for the entire duration of the study (i.e., through Week 52).

Exclusion Criteria

Subjects who met any of the following criteria were not eligible to participate in this study:

1. Weighed ≤50 kg (110 lbs) or ≥120 kg (265 lbs).
2. Were pregnant or breastfeeding or intended to conceive during the study period (i.e., through Week 52).
3. Received a stem cell transplant or a solid organ transplant other than a kidney transplant.
4. Had suspected CMV disease (either syndrome or tissue-invasive disease) or detectable CMV viremia by the central virology laboratory prior to the first dose of study drug.
5. Had a history of CMV disease (either syndrome or tissue-invasive disease) within 6 months prior to the first dose of study drug.
6. Had an absolute neutrophil count of <500 cells/μL, platelet count of <25,000/μL, or hemoglobin of <8 g/dL at screening.
7. Had hypersensitivity (not including renal dysfunction or an eye disorder) to valganciclovir (vGCV), ganciclovir (GCV), cidofovir (CDV) or to brincidofovir (BCV) or their excipients.
8. Received (or were anticipated to need treatment with) any of the following:

   * GCV, vGCV, foscarnet, intravenous CDV, or any other anti-CMV therapy (including CMV immune globulin, cell-based therapies, and investigational anti-CMV drugs, e.g., leflunomide, letermovir [previously AIC246], or maribavir) at any time posttransplant;
   * Any anti-CMV vaccine at any time;
   * Any other investigational drug within 14 days prior to the first dose of study drug (unless prior approval had been received from the Chimerix Medical Monitor or designee); or
   * Prior treatment with BCV at any time. [Note: An "investigational drug" was defined as any drug that is not approved for any indication by the FDA (or appropriate regulatory authority).]
9. Received acyclovir orally at >2000 mg total daily dose (TDD) or intravenously at >15 mg/kg TDD, valacyclovir at >3000 mg TDD on the first dose of study drug or were anticipated to receive any of these drugs at the doses described after the the first dose of study drug.
10. Were infected with HIV, hepatitis B virus (HBV), and/or hepatitis C virus (HCV), had evidence of active viral replication within 6 months prior to screening, as demonstrated by detectable HIV or HCV RNA, or detectable HBV DNA in blood, plasma or serum.
11. Had severe vomiting, diarrhea, or malabsorption syndrome on or prior to the first dose of study drug.
12. Had gastrointestinal (GI) disease that would have, in the judgement of the investigator, precluded the subject form taking or absorbing oral medication (e.g., gastroparesis, diabetic autonomic neuropathy affecting the GI tract, clinically active Crohn's disease, ischemic colitis, moderate or severe ulcerative colitis, small bowel resection, ileus, or any condition that was expected to require abdominal surgery during the course of study participation).
13. Had serum alanine aminotransferase or aspartate aminotransferase concentrations >5 x the upper limit of normal (ULN).
14. Had total serum bilirubin >2 x the ULN and direct bilirubin >1.5x the ULN.
15. Had moderate (Class B) to severe (Class C) hepatic dysfunction according to the Child-Pugh Turcotte scoring system.
16. Were receiving or would require digoxin or ketoconazole therapy (other than topical formulations) during the treatment phase of the study.
17. Had active malignancies (with the exception of basal cell carcinoma).
18. Had a serious psychiatric, medical disorder, including abnormal laboratory values, that would have, in the judgement of the investigator, put the subject at increased risk by participating in the study, or would have interfered with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - St. Vincent Medical Center, Los Angeles, California
  - University of Colorado Hospital/Health Science Center, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment 1 | Treatment 2
Started | 2 | 3
Completed | 0 | 0
Not Completed | 2 | 3
Not completed — Study Terminated | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Treatment 1: BCV plus vGCV placebo
  Brincidofovir
- Treatment 2: vGCV plus BCV placebo
  Valganciclovir
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 37 [27 to 47] | 44.3 [29 to 56] | 41 [27 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of CMV Disease
Description: The incidence of CMV disease included CMV tissue-invasive disease and CMV syndrome, occurring anytime between randomization and Week 52 (± 28 days).
  The proportion of subjects that met this failure endpoint were to be compared between brincidofovir (BCV) and valganciclovir (vGCV) using an unadjusted 95% confidence interval (CI) of the absolute difference between groups (BCV minus vGCV). If the upper bound of the 95% CI fell below 10%, BCV would have demonstrated non-inferiority to vGCV. In the event that the upper bound of the 95% CI fell below 0%, BCV would have additionally demonstrated superiority over vGCV.
Time Frame: 52 weeks (± 28 days)
Population: The study was terminated. Enrollment was suspended and all blinded study treatment was discontinued in early January 2016. Due to the premature termination of this study, statistical analyses were not performed. Limited demographic and safety data were provided for the 5 subjects enrolled.
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Treatment 1 | Treatment 2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=2) | Treatment 2 (N=3)
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Perinephric collection (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment 1 (N=2) | Treatment 2 (N=3)
Flatulence (Gastrointestinal disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
No conclusions regarding safety or efficacy can be made from the limited data obtained in this study. Enrollment was suspended and all blinded study treatment was discontinued early January 2016.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publications may be delayed up to an additional 90 days to allow Sponsor to seek patent protection.